CLINICAL TRIAL: NCT00586638
Title: Pilot Study Using a Video Game to Train Cognitive Control Processes in Healthy Older Adults
Brief Title: Training Cognitive Control Processes in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Yaakov Stern, Professor of Clinical, Department of Neurology Administration, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AAAC6151
Record Dates: First submitted 2007-12-20; First posted 2008-01-04 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Neurologic Manifestations; Neurobehavioral Manifestations
Keywords: cognition; cognition disorders; executive function; cognitive control; attentional control; biomedical enhancement; cognitive enhancement; computerized; computer-based; video game
MeSH Terms: conditions — Neurologic Manifestations; Neurobehavioral Manifestations; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Video Game play with training strategy
  Interventions: Behavioral: Video game based training
- 2 (Active Comparator): Video game play without training strategy
  Interventions: Behavioral: Video game based training
- 3 (No Intervention): Minimal contact control

INTERVENTIONS:
Behavioral: Video game based training — 36 one-hour sessions over 12 weeks
  Arms: 1; 2

SUMMARY:
Control processes are classes of brain activity that initiate, coordinate, synchronize, and regulate elemental cognitive functions for the conduct of goal-directed behavior. The proposed research investigates whether exposure to a computer-based training protocol designed to enhance cognitive control processes will improve cognitive performance in healthy older adults.

DETAILED DESCRIPTION:
The proposed research investigates whether exposure to a computer-based training protocol designed to enhance cognitive control processes will improve cognitive performance in healthy older adults. Cognitively normal adults aged 60-75 will be randomized into three experimental groups: 1) Video game play with training strategy; 2) Video game play without training strategy (Active Control); 3) Minimal contact (Passive Control). Subjects in Groups 1 and 2 will be instructed to play the complex, high-demand video game, Space Fortress, for 36 one-hour sessions over 12 weeks. Subjects in Group 3 will receive all assessments but will not play the computer game.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-75
* Willingness to adhere to training protocol
* Adequate English proficiency

Exclusion Criteria:

* Known history of cognitive impairment, dementia, stroke, seizure disorder, or other neuropsychiatric condition judged to impact cognitive performance
* Taking medications known to influence cognitive performance
* Sensory (e.g. visual, auditory) or physical (e.g. severe arthritic, orthopedic, neurologic) impairment incompatible with use of a standard computer workstation.
* Enrolled in a concurrent study that could affect the outcome of this study

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Neuropsychological testing | Week 1, 12, 24
Cognitive-experimental tasks | Week 1, 6, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Stern, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Result] Blumen HM, Gopher D, Steinerman JR, Stern Y. Training cognitive control in older adults with the space fortress game: the role of training instructions and basic motor ability. Front Aging Neurosci. 2010 Nov 11;2:145. doi: 10.3389/fnagi.2010.00145. eCollection 2010. PMID 21120135
- [Result] Stern Y, Blumen HM, Rich LW, Richards A, Herzberg G, Gopher D. Space Fortress game training and executive control in older adults: a pilot intervention. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2011 Nov;18(6):653-77. doi: 10.1080/13825585.2011.613450. Epub 2011 Oct 12. PMID 21988726